CLINICAL TRIAL: NCT02268188
Title: Harvesting Health for Cancer Survivors: A Pilot Project
Brief Title: Harvesting Health Program in Improving Diet and Physical Activity Level in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-14013; NCI-2014-01498 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Cancer Survivor
Keywords: Cancer Survivors
MeSH Terms: interventions — Educational Status; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (Harvesting Health program) (Experimental): Participants undergo a series of 10 education and training sessions over 1 hour every 2 weeks, comprising education on current research, evidence-based health guidelines, application techniques, reference materials specific to extended-stage cancer survivors, and recommendations and personal health goals for survivorship. The guidelines described in class are part of a nutrition intervention and an exercise intervention with personal and group goal setting over the course of the study.
  Interventions: Other: education; Other: nutrition intervention; Behavioral: exercise intervention; Other: questionnaire administration; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Other: education — Attend classes as part of Harvesting Health program
Other: nutrition intervention — Learn how to incorporate nutrition guidelines into daily meal plans as part of Harvesting Health program
Behavioral: exercise intervention — Use FitBit to log daily steps as part of Harvesting Health program
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies the Harvesting Health Program in improving the diet and physical activity level of cancer survivors. Nutrition and physical activity classes and the opportunity to harvest fruits, vegetables, and herbs may increase participants' fruit and vegetable consumption and physical activity levels. Studying the participation rates and changes in participants' eating and physical activity habits may help doctors learn whether the program has an effect on participant lifestyle.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure survivor participation in regards to each aspect of the Harvesting Health Program (personalized and group education, gardening and harvesting, and utilization of novel web-based technologies).

II. Assess survivor preferences regarding key Harvesting Health Program components impacting participation (physical facilities, schedule and timing, education topics and sessions, garden access, web portal usability, etc.).

SECONDARY OBJECTIVES:

I. A customized "Nutrition & Physical Activity Scorecard" has been developed and will be implemented to evaluate pre/post measures of diet and physical activity at baseline (month 0) and at months 6, 9 and 12.

II. Participants are evaluated at baseline and at completion of the intervention for: (a) serum and body composition biomarkers of exposure and efficacy, and (b) health indices related to cancer survivorship and overall health.

III. To assess Program sustainability, follow-up questionnaires will be completed at 9 and 12 months using the Nutrition & Physical Activity Scorecard and questionnaires regarding quality of life outcomes.

OUTLINE:

Participants undergo a series of 10 education and training sessions over 1 hour every 2 weeks, comprising education on current research, evidence-based health guidelines, application techniques, reference materials specific to extended-stage cancer survivors, and recommendations and personal health goals for survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to participate and sign an informed consent document
* Adults with the ability to read, write, and speak English who have access to the internet
* Cancer survivors who have completed active cancer treatments within the previous 12 months extended-stage survivors)
* Survivors must have a computer with internet access and an active email account
* Participants must refrain from traveling for more than 3 weeks total during the intervention period
* Participants who are undergoing long-term hormone therapy (i.e., tamoxifen) are permitted to enroll

Exclusion Criteria:

* Cancer survivors who are cognitively unable to consent or have physical or mental limitations that would prevent full participation in the program
* Adults receiving active treatment including surgery, neoadjuvant hormonal, chemotherapy, or radiation
* Survivors with pre-existing medical conditions that preclude unsupervised physical activity (i.e., severe orthopedic conditions, impending hip or knee replacement, paralysis, unstable angina, dementia, or recent history of myocardial infarction, congestive heart failure, pulmonary conditions that require oxygen, or hospitalization within six months)
* Adults taking any medication that do not allow for increased intake of fruits and vegetables (i.e., pharmacologic doses of warfarin)
* Survivors currently involved in other clinical trials
* Long-term cancer survivors (> 12 months post treatment)
* Those planning to start certain medications after the trial enrollment or use of non- prescription substances (i.e. saw palmetto and other herbal or alternative products)
* Survivors with active metabolic or digestive illnesses such as malabsorptive disorders (Crohn's, celiac disease, irritable bowel syndrome [IBS]), renal insufficiency, hepatic insufficiency, cachexia, or short bowel syndrome
* Pregnant women will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of sessions attended, as measured by mobile scanner | Up to 6 months
  Analyzed with standard descriptive statistics. Measures of central tendency (mean and/or median) and spread (standard deviation, quartiles, minimum and maximum) will be reported.
Number of hits on the web portal | Up to 12 months
  Analyzed with standard descriptive statistics. Measures of central tendency (mean and/or median) and spread (standard deviation, quartiles, minimum and maximum) will be reported.

SECONDARY OUTCOMES:
Number of web hits on portal pages | Up to 12 months
  Quantitative and qualitative analysis will be performed on the harvest log to determine common themes and feedback from the participants.
Program evaluation overall score | Up to 20 weeks
  Quantitative and qualitative analysis will be performed on the harvest log to determine common themes and feedback from the participants.
Change in behavior, measured by Nutrition & Physical Activity Scorecards | Baseline to 12 months
  The hypothesis of no change in the overall scorecard value will be tested versus a two sided alternative using a paired T-test at alpha level 0.025 (Bonferroni corrected for 2 scorecards). Exploratory analyses may be completed to understand which components of these Scorecards are driving the improvement or degradation in scores.
Change in biomarker levels, assessed by values for the Health & Wellness Index | Baseline to 6 months
  Biomarkers include blood glucose, lipid panel (total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides), skin antioxidant score and bone density. The hypothesis of no change in these markers will be tested using a multivariate Hotelling's T-squared test at the 0.05 level. If a significant difference is noted, then the individual scores will be further tested with paired t-tests to determine which are significantly different. The p-values of the individual t-tests will be adjusted via a Bonferroni correction.
Change in physical activity using the International Physical Activity Questionnaire | Baseline to 12 months
  This questionnaire categorizes respondents into "Low", "Moderate", or "High" activity levels based upon survey responses.
Change in nutrient intake | Baseline to 6 months
  Viowell food frequency questionnaire

OTHER OUTCOMES:
Change in Quality of Life using the Short Form-12 (SF-12) | Baseline to 6 months
  The SF-12 is a
Change in depression scale using the Center for Epidemiologic Studies Depression Scale Revised (CED-R) | Baseline to 6 months
  The CED-R is a screening test for depression and depressive disorder. The range of scores is between 0 and 60 and a score over 16 indicates depression.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Spees CK, Braun AC, Hill EB, Grainger EM, Portner J, Young GS, Kleinhenz MD, Chitchumroonchokchai C, Clinton SK. Impact of a Tailored Nutrition and Lifestyle Intervention for Overweight Cancer Survivors on Dietary Patterns, Physical Activity, Quality of Life, and Cardiometabolic Profiles. J Oncol. 2019 Nov 21;2019:1503195. doi: 10.1155/2019/1503195. eCollection 2019. PMID 31871455
- See also: The Jamesline — http://cancer.osu.edu